CLINICAL TRIAL: NCT00220896
Title: Prevention of Postoperative Delirium With Donepezil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Eisai Deutschland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PSYTUM1
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Cognitively Normal Elderly Individuals
Keywords: Delirium; Prevention; Donepezil
MeSH Terms: conditions — Delirium | interventions — Donepezil

INTERVENTIONS:
Drug: Donepezil

SUMMARY:
Patients undergoing hip or knee joint replacement at the age of 70 years or above who are cognitively unimpaired will receive donepezil or matching placebo before (over 5-7 days), during and after (over 7 days) surgery. The incidence of delirium will be monitored at 3 days, 7 days, and 49 days following surgery. We hypothesize that the incidence of delirium can be lowered from 20 per cent to 10 per cent by the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively healthy, elective hip or knee replacement

Exclusion Criteria:

* Ongoing cholinergic treatment, dementia, delirium, acute physical illness

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-01; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium

SECONDARY OUTCOMES:
Cognitive performance

CONTACTS AND LOCATIONS:
Overall Officials: Janine Diehl, M. D., Principal Investigator — Dept. of Psychiatry, Technische Universitaet Muenchen
Locations (1):
- Deps. of Psychiatry and Anaesthesiology, Tech. Universitaet Munich, Munich, Germany